CLINICAL TRIAL: NCT03446898
Title: A Cohort Study of the Effect of High Altitudes on Physiological and Metabolic Markers in Adults Who Live at Qinghai-Tibet Plateau for Work Purpose
Brief Title: A Study of the Effect of High Altitudes on Physiological and Metabolic Markers in Adults Living at Qinghai-Tibet Plateau for Work Purpose
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tibetan Traditional Medical College (Other)
Collaborators: Beijing University of Chinese Medicine (Other); Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: Z2016B01G03/02-CRP
Record Dates: First submitted 2018-01-30; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Residence or Prolonged Visit at High Altitude as the Cause of Mountain Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults Living at Qinghai-Tibet Plateau for Work Purpose: Qinghai-Tibet Plateau is a high altitude area in which human would be exposed in chronic hypoxia environment.
  Interventions: Other: Chronic hypoxic environment

INTERVENTIONS:
Other: Chronic hypoxic environment — Chronic hypoxic environment. Since the partial pressure of oxygen in inspired air falls with increasing terrestrial elevation above sea level, many physiological variables in adults would be affected by the chronic hypoxia environment.

SUMMARY:
This ambispective cohort study aims to evaluate the effect of high altitudes environment on human's physiological and metabolic markers, specific markers of main human systems, and incidence rate and severity of chronic mountain sickness (CMS).

DETAILED DESCRIPTION:
Qinghai-Tibet plateau is a high altitudes area with average 3,000-5,000 meters height in China. As the partial pressure of oxygen in inspired air falls with increasing terrestrial elevation above sea level, many physiological variables in human body could be affected by this hypobaric hypoxic environment. Up to date, there are no large scale clinical trials assessing these changes in chinese population. The study here would like to provide the newest medical information on the changes of physiological variables and correlation between specific risk factors in chinese adults living at high altitudes for work purpose.

ELIGIBILITY:
Inclusion Criteria:

* Be provided verbal or written informed consent;
* Men and women ≥ 30 and ≤ 65 years of age;
* Adults living at Qinghai-Tibet Plateau for Work Purpose, and the altitude of residence is more than 2,500 meters;
* Providing electronical or paper medical examination reports which conducted in 2016.

Exclusion Criteria:

* Pregnant or breast-feeding women;
* Be excluded by Principal investigator for subject's compliance or safety reasons.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is adults who live at Qinghai-Tibet Plateau for Work Purpose.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2017-07-22 (Actual); Primary Completion 2018-03-22 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in weight from baseline at first year | Baseline and 1st year
Change in blood pressure as measured by sphygmomanometer from baseline at first year | Baseline and 1st year
  The blood pressure will be described in the format of diastolic pressure/systolic pressure, and the unit of measure is mmHg.
Change in serum lipid from baseline at first year | Baseline and 1st year
Change in blood glucose from baseline at first year | Baseline and 1st year

SECONDARY OUTCOMES:
Change in weight from baseline at second year | Baseline and 2nd year
Change in weight from baseline at third year | Baseline and 3rd year
Change in blood pressure as measured by sphygmomanometer from baseline at second year | Baseline and 2nd year
  The blood pressure will be described in the format of diastolic pressure/systolic pressure, and the unit of measure is mmHg.
Change in blood pressure as measured by sphygmomanometer from baseline at third year | Baseline and 3rd year
  The blood pressure will be described in the format of diastolic pressure/systolic pressure, and the unit of measure is mmHg.
Change in serum lipid from baseline at second year | Baseline and 2nd year
Change in serum lipid from baseline at third year | Baseline and 3rd year
Change in blood glucose from baseline at second year | Baseline and 2nd year
Change in blood glucose from baseline at third year | Baseline and 3rd year
Pathological changes from baseline at first year in human body systems | Baseline and 1st year
Pathological changes from baseline at second year in human body systems | Baseline and 2nd year
Pathological changes from baseline at third year in human body systems | Baseline and 3rd year
The incidence rate and severity of chronic mountain sickness (CMS) | The 2nd year
  The diagnosis and severity of CMS is identified and assessed using "The Qinghai Chronic Mountain Sickness Score". The score ranges from 0 to 27, and a higher value means a worse outcome.
The incidence rate and severity of chronic mountain sickness (CMS) | The 3rd year
  The diagnosis and severity of CMS is identified and assessed using "The Qinghai Chronic Mountain Sickness Score". The score ranges from 0 to 27, and a higher value means a worse outcome.

OTHER OUTCOMES:
Relationship between altitudes and pathological changes in human body under chronic hypoxic environment | Up to the 3rd year
Relationship between age and pathological changes in human body under chronic hypoxic environment | Up to the 3rd year
Relationship between gender and pathological changes in human body under chronic hypoxic environment | Up to the 3rd year

CONTACTS AND LOCATIONS:
Overall Officials: Tonghua Liu, Professor, Principal Investigator — Tibetan Traditional Medical College
Locations (1):
- Tibetan Traditional Medical College, Lhasa, Tibet, China

IPD SHARING:
Plan to Share IPD: Undecided